CLINICAL TRIAL: NCT03649646
Title: A Multi-center, Open, Longitudinal, Observational Study to Assess the Treatment Trend and the Proportion of Target BP Attainment in Patients Whose Antihypertensive Regimens Are Changed to ARB-based Therapy
Brief Title: FimasaRtan-basEd BP Targets After Drug SwitcHing
Acronym: FRESH
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-404
Record Dates: First submitted 2018-08-08; First posted 2018-08-28 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2018-08

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Fimasartan
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with hypertension uncontrolled by antihypertensive drug

SUMMARY:
The recent hypertension clinical practice guidelines published by American College of Cardiology (ACC) and American Heart Association (AHA) reduced the target BP to 130/80 mmHg, indicating the needs for more aggressive efforts in hypertension treatment. However, studies in Koreans must be preceded before applying such new overseas guidelines; thus, this study has been designed to establish clinical materials reflecting treatment setting in Korea. In this study, patients with uncontrolled hypertension whose antihypertensive regimens are changed to ARB-based therapy (ARB monotherapy or ARB-containing combination therapy) will be followed to assess the treatment trend, treatment effect, and risk of cardiovascular disease.

DETAILED DESCRIPTION:
This study will be performed in patients with blood pressure (BP) uncontrolled by existing antihypertensive drugs (including ARB) among hypertensive patients visiting outpatient clinic of medical institutions in Korea. The study enrollment number will be assigned to the subjects who provide a written consent to the use of personal information and meet the inclusion/exclusion criteria. Follow-up will be conducted for 12 weeks in total and prespecified study related data will be collected in the case report form.

ELIGIBILITY:
Inclusion Criteria:

* Provided written consent to the use of personal information after receiving the explanation of the objective, methodology, etc. of this clinical study
* Male or female adults ≥ 19 years who are diagnosed with essential hypertension
* Receiving outpatient treatment at the time of study enrollment
* Patients with hypertension uncontrolled by existing antihypertensive drugs (including ARB) whose antihypertensive regimens decided and scheduled to be changed to ARB monotherapy or ARB-containing combination therapy (the result of the arm with a higher mean BP [systolic BP preferred] when measured twice with at least a 2-minute interval in both arms at the medical office on the study enrollment date, will become the reference)

  * Definition of uncontrolled hypertension: Target BP (SBP <140 mmHg and DBP <90 mmHg) not achieved even after the treatment using the existing antihypertensive drugs for 4 weeks or longer

Exclusion Criteria:

* Patients who were hospitalized or are scheduled to be hospitalized 4 weeks before or after the study enrollment date
* Patients with suspected or confirmed secondary hypertension
* Pregnant or breast-feeding women
* Patients who received investigational product within 12 weeks or are scheduled to participate in another clinical study while participating in this study
* Patients who are determined inappropriate for participating in the study by investigators for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension uncontrolled by antihypertensive drugs* whose antihypertensive regimens are changed to angiotensin receptor blocker (ARB) monotherapy or concomitant antihypertensive drug therapy containing ARB.
  *Including patients who previously received angiotensin receptor blocker (ARB); in this case, changing to other therapy using an ARB with different ingredient is allowed.
Sampling Method: Non-Probability Sample
Enrollment: 4542 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Ajou University Hospital, Suwon, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 4542
Completed | 4075
Not Completed | 467

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 4075
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.63 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2184
  Male | 1891
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 4075
BMI [Mean (Standard Deviation); unit: kg/㎡] | 25.33 (3.36)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Controlled Blood Pressure (<140/90 mmHg)
Description: Percentage of patients who attain the target blood pressure (BP) (<140(SBP)/90(DBP) mmHg) at Week 12 after the treatment regimen change
Time Frame: Week 12 after the treatment regimen change
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 4075
Participants | 3083

2. Secondary Outcome: Percentage of Patients With Controlled BP According to 2018 KSH Guideline
Description: Percentage of patients who attain the target BP specified in 2018 hypertension clinical practice guidelines* suggested by Korean Society of Hypertension at Week 12 after the treatment regimen change.
  *2018 hypertension clinical practice guidelines : Target BP <140(SBP)/90(DBP) mmHg.
  For patients meeting any of the conditions listed below, each corresponding criterion will be applied.
  * Patients with cardiovascular disease :<130/80 mmHg
  * Patients with diabetes : <140/85 mmHg
  * Patients with diabetes accompanying cardiovascular disease :<130/80 mmHg
  * Patients with chronic kidney disease accompanying albuminuria: <130/80 mmHg
Time Frame: Week 12 after the treatment regimen change
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 4075
Participants | 2353

3. Secondary Outcome: Percentage of Patients With Controlled BP According to 2017 ACC/AHA Guideline
Description: Percentage of patients who attain the target BP(<130(SBP)/80(DBP)mmHg) specified in 2017 clinical practice guidelines for hypertension suggested by American College of Cardiology(ACC)/American Heart Association(AHA) at Week 12 after the treatment regimen change
Time Frame: Week 12 after the treatment regimen change
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 4075
Participants | 1454

4. Secondary Outcome: Prcentage of Patients With Controlled BP According to Investigator's Target BP
Description: Percentage of patients who attain the investigator's target BP* at Week 12 after the treatment regimen change.
  *Investigator's target BP: Target BP for each patient set by the investigator at baseline.
Time Frame: Week 12 after the treatment regimen change
Population: Missing of investigator's target BP: 4 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Patients
Number analyzed (Participants) | 4071
Participants | 1388

ADVERSE EVENTS:
Time Frame: Week 12
Description: SAEs and antihypertensive drug related ADRs were collected during the study period.
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 2/4386
Serious Adverse Events (participants affected / at risk) | 18/4386
Other Adverse Events (participants affected / at risk) | 37/4386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=4386)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=4386)
Palpitations (Cardiac disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Dizziness postural (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 13 (13)
Headache (Nervous system disorders) | 5 (5)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT03649646/Prot_SAP_000.pdf